CLINICAL TRIAL: NCT03150745
Title: Office Hysteroscopy Versus Stationary Coloposcopy for Diagnosis of Cervical Lesions in Women With Unhealthy Looking Cervix
Brief Title: Diagnosis of Cervical Lesions in Women With Unhealthy Looking Cervix
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Lecturer of obstetrics and gynecology, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CLLC
Record Dates: First submitted 2017-05-09; First posted 2017-05-12 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Cervical Dysplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Colposcopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colposcopic group (Other)
  Interventions: Procedure: 3- Cervical Pap smears; Procedure: Colposcopic examination
- office hysteroscopic group (Other)
  Interventions: Procedure: 3- Cervical Pap smears; Procedure: Office hysteroscopy

INTERVENTIONS:
Procedure: 3- Cervical Pap smears — Cervical Pap smears will be obtained using the long tip of an Ayre's spatula that will be placed in the endocervical canal with the proximal bulge resting on the ectocervix. The spatula will be carefully rotated around the cervix so that a representative sample of the whole cervix will be obtained. An additional endocervical sample will be obtained by placing a cytobrush or by the other end of the Ayer's spatula in the endocervical canal and gently rotated through 360 degrees as previously described. The samples will be then immediately plated on a slide, fixed by immersing the slide in 95% ethyl alcohol fixative for 15 to 20 minutes and stained by modified Papanicolaou stain using a hand staining procedure
Procedure: Colposcopic examination — 0.9% saline technique to assess the cervical lesion and vasculature of the cervix, 5% acetic acid technique to determine acetowhite-positive areas. Schiller's iodine technique to visualize high glycogen containing cells. Endocervical canal assessment using (Bossman forceps or endocervical speculum or counter pressure with Q stick).
  e- Biopsy using the punch biopsy forceps. Biopsy will be obtained from every abnormal colposcopic examination
  Arms: Colposcopic group
Procedure: Office hysteroscopy — 0.9% saline technique to assess the cervical lesion and vasculature of the cervix. 5% acetic acid technique to determine acetowhite-positive areas. Schiller's iodine technique to visualize high glycogen containing cells. Endocervical canal assessment. Endometrial cavity evaluation whenever possible. Biopsy. Biopsy will be obtained from every abnormal hysteroscopic examination.
  Arms: office hysteroscopic group

SUMMARY:
Endocervix (cervical canal) is the cavity of the cervix and connects the external os with the internal os. It is fusiform in shape and has posterior and anterior oblique longitudinal ridges, the plicae palmatae. These are not exactly apposed but inter-lock like a zipper so that the canal is kept closed.

The original squamous epithelium is clearly identified as a smooth, usually featureless covering of the cervix; its uniform pink color contrasts with the redness of the original columnar epithelium. It joins the latter at the original squamocolumnar junction.

Many clinicians encounter cervical lesions that may or may not be associated with cytologic abnormalities. Such abnormalities as ectropion, Nabothian cysts, and small cervical polyps are quite benign and need not generate concern for patient or clinician, whereas others, including those associated with a history of exposure to diethylstilbestrol, cervical inflammation, abnormal cervical cytology, and postcoital bleeding, should prompt additional evaluation. Further, in some patients, the cervix may be difficult to visualize. Several useful clinical suggestions for the optimal examination of the cervix are presented.

ELIGIBILITY:
Inclusion Criteria:

1. Suspicious cervix
2. Age between 20 to 60 years

Exclusion Criteria:

1. Previously diagnosed cervical lesions.
2. Pregnant women.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
The sensitivity of office hysteroscopy detection of cervical lesions | 1 week
The sensitivity of colposcopy | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided